CLINICAL TRIAL: NCT00727948
Title: The Impact of the Anti-Platelet Agent Aspirin on Angiogenesis Proteins in Women With Breast Cancer
Brief Title: The Effect of Aspirin on Angiogenesis Proteins in Women on Tamoxifen Therapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Chris Holmes, Associate Professor of Medicine, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V0801
Record Dates: First submitted 2008-07-30; First posted 2008-08-04 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2010-06

CONDITIONS: Breast Cancer; Angiogenesis
Keywords: Breast cancer; Angiogenesis; Aspirin; Tamoxifen
MeSH Terms: conditions — Breast Neoplasms | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- receive aspirin (Experimental)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — 325 mg tablets, once daily for 45 days

SUMMARY:
Changes in major angiogenic proteins have been seen following initiation of tamoxifen and aromatase inhibitor therapy in women with breast cancer. One source of these proteins is the circulating platelet pool. The investigators hypothesize that in addition to their anti-platelet properties, agents such as aspirin can be used as targeted anti-angiogenesis therapy. The investigators will determine the influence of aspirin on the release of angiogenic proteins from platelets in 35 patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven breast cancer
* Pre or post-menopausal
* Age >18
* Completed adjuvant non-hormonal therapy >30 days prior to initiation of study (surgery and/or chemotherapy and/or radiation therapy)
* Platelet count and hemoglobin within normal ranges for local lab within 30 days of initiation of study therapy
* Receiving tamoxifen therapy for at least 90 days prior to initiation of study therapy, and is expected to continue that therapy for the duration of the study (75 days)

Exclusion Criteria:

* Chemotherapy, radiation therapy or surgery within 30 days of study therapy
* Current use of aspirin, anti-platelet or anti-coagulation agents on a continuous basis
* Prior history of gastrointestinal or central nervous system bleeding, or documented or self-reported blood in stools or bright red blood per rectum

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes in pro-angiogenic and anti-angiogenic protein levels. | 75 days

CONTACTS AND LOCATIONS:
Overall Officials: Chris E Holmes, MD, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States